CLINICAL TRIAL: NCT03904771
Title: Food for Mind - Group-based Behavioral Nutrition Intervention in the Treatment of Depression
Brief Title: Food for Mind - Intervention in the Treatment of Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Eastern Finland (Other)
Collaborators: Social Insurance Institution, Finland (Other); Finnish Cultural Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FoMi
Record Dates: First submitted 2018-12-19; First posted 2019-04-05 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food for Mind -intervention group (Active Comparator): Nutrition counselling + peer support
  Interventions: Behavioral: Nutrition counselling + peer support
- Befriending group -control group (Active Comparator): Social activation + peer support
  Interventions: Behavioral: Social activation + peer support

INTERVENTIONS:
Behavioral: Nutrition counselling + peer support — Behavioral nutrition counselling and peer support, delivered in small groups. Includes six sessions extending over 8 weeks, with participatory activities facilitated by a nutrition therapist.
  Arms: Food for Mind -intervention group
Behavioral: Social activation + peer support — Social activation and peer support, delivered in small groups. Includes six sessions extending over 8 weeks, with participatory activities facilitated by group leader.
  Arms: Befriending group -control group

SUMMARY:
Aims. The main aim of the study is to explore whether Food for Mind - Group-based behavioral nutrition intervention alleviates depression symptoms. Furthermore, we aim to investigate, whether the intervention improves the quality of diet, eating habits, quality of life, ability to work and to study its cost-effectiveness.

In collaboration with 11 public and private health care service providers in cities of Kuopio and Siilinjärvi in Northern Savo, Finland.

Participants. The total number of subjects will be 144 based on power calculations. The calculation is based on the clinical decline of seven points assessed by the Center for Epidemiologic Studies Depression (CES-D) Scale. Participants sign an informed consent form to participate Food for Mind - intervention.

Study design.

In this randomized controlled clinical trial subjects are randomized into two parallel groups: Food for Mind -behavioral nutrition intervention group (n=72) and Group to bring Good Mood -control group (n=72).

The intervention consists of behavioral nutrition counselling (5 times 1½ h and 1 time 3 h) and the control group (befriending group) (n=72) (5 times 1½ h and 1 time 3 h). Thus, in the befriending group the same visit schedule and length without any nutrition counselling is used. The befriending group consists of discussion of neutral topics, like hobbies, music, sports, and doing together. Both groups continue to have their normal depression care in the health care.

Enrollment and treatment will take about four years, and follow-up will last about one year.

The Northern Savo Hospital District Committee on Research Ethics gave its consent to the study protocol.

Methods. All questionnaires are validated. CES-D -depression scale, Seasonal Pattern Assessment Questionnaire, The Diet Quality Index (IDQ), Diet frequency -questionnaire, Eating competence -questionnaire (ecSI 2.0), The Three Factor Eating Questionnaire, Ability to work and function -questionnaires, Assessment of Quality of Life (AQoL)-8D (8 dimensions) -questionnaire, Treatment expectancy -questionnaire, Acceptability -questioinnaire.

In addition, body composition measurement and cost-effectiveness analyses to evaluate the health outcomes in relation to resource utilization and costs in Food for Mind -intervention.

DETAILED DESCRIPTION:
Food for Mind -intervention group - topics of small group meetings

1. Getting to know each other and forming a group.
2. Overall quality of diet and meal rhythm, shifting thoughts to changing of wishes.
3. Nutrition and depression based on the evidence based studies
4. Mindful Eating - practical Food for Mind cooking class and eating meal together applying mindful eating
5. Food for Mind - getting to know a selection of Food for Mind -food items available in the grocery store.
6. Tools for the future: discovering and ensuring your own tools for success to put into action.

Participants in the Food for Mind -intervention group will get for every group meeting optional home exercises consisting of observing their own food habits and bringing "food for mind" items on their meal plan. As a social support, participants can share their own experiences and findings via WhatsApp (Whats Application) messenger -mobile application. The WhatsApp messenger-mobile application is used during the intervention and ten months after it.

The behavioral nutrition counselling is theory-based, i.e. solution focused theory (SFT) and self -determination theory. SFT places responsibility for change in the hands of subjects by using empowering language and recognizing them as skilled in matters of self-care. Subjects have strengths, resources, and coping skills that drive change while generating optimism and hope. Use of basic counseling skills, such as attending and listening, genuineness, empathy, positive regard and reflection, provide the foundation upon which SFT is practised.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 - 65 years
2. Customer Relationship of Kuopio Psychiatric Center or City of Kuopio: Individually tailored treatment and rehabilitation plan
3. ICD-10 (International Classification of Diseases 10th Revision): Depression Diagnosis (F32-F33, F34.1)
4. The treatment (medication and / or psychotherapy) has continued unchanged for at least 2 weeks time before randomization
5. Willingness to participate in group-based intervention for 8 weeks: 6 group sessions (5 x 1½h and 1 x 3h)

Exclusion Criteria:

1. General illness that is clinically unstable and which can be aggravated by intervention
2. Pregnancy
3. Severe food allergy, intolerance or food aversion
4. Participation at the same time, such as other nutrition or exercise intervention
5. Primary diagnosis include personality disorder, severe eating disorder and / or substance abuse.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Depressive Symptomatology at eight weeks, 6 months and 12 months. | 12 months: assessed at baseline, at eight weeks, at 6 months and at 12 months.
  Depressive symptomatology measured with the Center for Epidemiologic Studies (CES-D) scale at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
  The scale has 20 items and measures symptoms of depression. Each item is scored from 0 (zero) to 3 points. The total score ranges from 0 (zero) to 60 points.Higher values of the total score represent a worse outcome.Four of the items (#4, #8, #12, #16) are reversed before calculating the total score. The total score is calculated as follows: the answers to the items are summed, the sum is divided by the number of scored items, and this value is multiplied by 20. If the answers are missing to more than five items, the total score will not be calculated.

SECONDARY OUTCOMES:
Change from baseline Diet Quality at eight weeks, 6 months and 12 months. | 12 months: assessed at baseline, at eight weeks, at 6 months and at 12 months.
  The Diet Quality measured with the Diet Quality Index (IDQ) at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
Change from baseline Diet Frequency at eight weeks, 6 months and 12 months. | 12 months: assessed at baseline, at eight weeks, at 6 months and at 12 months.
  The Diet Frequency measured with the Diet frequency -questionnaire at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
Change from baseline Eating Competence at eight weeks, 6 months and 12 months. | 12 months: assessed at baseline, at eight weeks, at 6 months and at 12 months.
  Eating Competence measured with the Eating competence -questionnaire (ecSI 2.0) at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
Change from baseline Eating Behavior at eight weeks, 6 months and 12 months. | 12 months: assessed at baseline, at eight weeks, at 6 months and at 12 months.
  Eating Behavior measured with The Three Factor Eating Questionnaire at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
Change from baseline Ability to Work and Function at eight weeks, 6 months and 12 months. | 12 months: assessed at baseline, at eight weeks, at 6 months and at 12 months.
  Ability to Work and Function measured with the Ability to work and function -questionnaires at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
Change from baseline Quality of Life at eight weeks, 6 months and 12 months. | 12 months: assessed at baseline, at eight weeks, at 6 months and at 12 months.
  The Quality of Life measured with the AQoL-8D -questionnaire at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.

OTHER OUTCOMES:
Change from baseline body weight at eight weeks, 6 months and 12 months. | 12 months: measured at baseline, at eight weeks, at 6 months and at 12 months.
  Body weight measured by body composition analyzer (InBody720) at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
Change from baseline fat mass at eight weeks, 6 months and 12 months. | 12 months: measured at baseline, at eight weeks, at 6 months and at 12 months.
  Fat mass measured by body composition analyzer (InBody720) at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.
Change from baseline fat free mass at eight weeks, 6 months and 12 months. | 12 months: measured at baseline, at eight weeks, at 6 months and at 12 months.
  Fat free mass measured by body composition analyzer (InBody720) at eight weeks, 6 months and 12 months after patient recruitment compared to the social support befriending group.

CONTACTS AND LOCATIONS:
Overall Officials: Outi M Nuutinen, PhD, Principal Investigator — Visiting researcher at the unit of Clinical Nutrition, UEF
Locations (1):
- Psychiatric Centre of Kuopio, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roponen J, Ruusunen A, Absetz P, Partonen T, Kuvaja-Kollner V, Hujo M, Nuutinen O. Nutrition-focused group intervention with a strength-based counseling approach for people with clinical depression: a study protocol for the Food for Mind randomized controlled trial. Trials. 2021 May 17;22(1):344. doi: 10.1186/s13063-021-05279-5. PMID 34001230